CLINICAL TRIAL: NCT06153810
Title: Efficacy of AesyBite Active in Reducing Sleep Bruxism Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesyra SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABA020-CIP-001
Record Dates: First submitted 2023-11-16; First posted 2023-12-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-01

CONDITIONS: Sleep Bruxism
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early stimulation (Experimental): Biofeedback treatment is started after two weeks of observation
  Interventions: Device: Biofeedback stimulation
- Delayed stimulation (Experimental): Biofeedback treatment is started after three weeks of observation
  Interventions: Device: Biofeedback stimulation

INTERVENTIONS:
Device: Biofeedback stimulation — Delivery of the vibratory biofeedback stimulus

SUMMARY:
The overall objective of the clinical investigation is to evaluate whether the use of the AesyBite Active reduces the bruxism activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years, in good general health.
* Presence of at least one of the following:

  * sleeping partner's report of tooth grinding sounds during sleep for at least three nights per week within the last 6 months,
  * hypertrophy of the masseter muscle upon digital palpation.
* Presence of at least one of the following:

  * signs of tooth attrition or shiny spots on dental restorations,
  * self-report of masticatory muscle fatigue or pain at awakening.
* Previous prescription of a night splint for bruxism.
* Able to understand and follow the protocol and complete the self-administered paper questionnaires.
* Able to provide written informed consent to study participation and storage and processing of study data

Exclusion Criteria:

* Allergic to Ethylene-Vinyl Acetate (EVA) copolymer.
* With more than two missing molars (excluding third molars).
* Ongoing orthodontic treatment (e.g. teeth alignment).
* With major neurological or psychiatric disorders including substance dependence.
* Using a removable dental prosthesis.
* Using a medication with known effects on sleep or motor behavior.
* Suffering from periodontal disease.
* With occlusal or jaw abnormalities that prevent the wearing of a normal dental splint.
* Participants with pacemakers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Reduction of the bruxism activity | 1 month
  Evaluation of the efficacy of AesyBite Active in reducing the bruxism activity expressed as total sleep bruxism duration per hour (TDPH, sec/hour) by at least 60% in the stimulation phase compared with baseline with a 10% non-inferiority margin.

SECONDARY OUTCOMES:
Reduction of the bruxism index | 1 month
  Evaluation of the efficacy of AesyBite Active in reducing the bruxism index expressed as number of sleep bruxism episodes per hour (episodes/hour).
Reduction of the mean duration of sleep bruxism episode | 1 month
  Evaluation of the efficacy of AesyBite Active in reducing the mean duration of sleep bruxism episodes (sec/episode).
Relative change in average intensity of bruxism episodes | 1 month
  A measure of the average bite strength exerted during the bruxism episodes.
Change in self-reported sleep quality marked on a visual analogue scale | 1 month
  Change in self-reported sleep quality assessed using a visual analogue scale (VAS) with a sleep quality scale from 0 to 10.
Change in self-reported pain marked on a visual analogue scale | 1 month
  Change in self-reported pain (facial pain, myofascial headache) assessed using a visual analogue scale (VAS) with a pain severity scale from 0 to 10.
Change in self-reported comfort marked on a visual analogue scale | 1 month
  Change in self-reported comfort assessed using a visual analogue scale (VAS) with a comfort severity scale from 0 to 10.
Change in self-reported retention marked on a visual analogue scale | 1 month
  Change in self-reported retention assessed using a visual analogue scale (VAS) with a retention severity scale from 0 to 10.
Change in self-reported ease of breathing marked on a visual analogue scale | 1 month
  Change in self-reported ease of breathing assessed using a visual analogue scale (VAS) with a ease of breathing severity scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Maddalone, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori
Locations (1):
- Fondazione Irccs San Gerardo Dei Tintori, Monza, Monza E Brianza, Italy